CLINICAL TRIAL: NCT03027115
Title: Post-operative Urinary Retention: A Prospective Randomized Study Identifying Patients at Risk and Reducing the Incidence Using Tamsulosin Pretreatment
Brief Title: Hernia Surgery Urinary Retention
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Health University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHUMC 2016.10.05
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Hernia; Urinary Retention
MeSH Terms: conditions — Hernia; Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: Randomization to 1 of 2 possible arms, control and treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): treatment with a selective alpha1-adrenoceptor antagonist
  Interventions: Drug: Tamsulosin
- Control (No Intervention): no treatment

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin treatment for 7 days pre-operatively
  Other Names: Flomax
  Arms: Treatment

SUMMARY:
Investigating whether pre-operative treatment with a selective alpha1-adrenoceptor antagonist affects the likelihood of male patients developing post-operative urinary retention following hernia repair.

DETAILED DESCRIPTION:
The purpose of this study will be to investigate whether pre-operative treatment with a selective alpha1-adrenoceptor antagonist affects the likelihood of male patients developing post-operative urinary retention following hernia repair surgery. It is also of interest to determine whether or not a well-known urological screening tool, the IPSS, can identify patients at risk for urinary retention following elective laparoscopic or open hernia repair surgery. We will investigate if it is possible to pre-treat patients with a selective alpha1-adrenoceptor antagonist which we think can reduce the incidence of post-operative urinary retention and the associated adverse consequences, especially in those patients at higher risk.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years of age
* Presenting with hernia requiring surgical intervention

Exclusion Criteria:

* Intolerability of tamsulosin or related drugs
* Investigator discretion
* Unwillingness or inability to comply with protocol procedures and assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-01-13 (Estimated); Study Completion 2020-01-27 (Estimated)

PRIMARY OUTCOMES:
Post-operative urinary retention | 2 weeks
  Incidence of post-operative urinary retention in patients undergoing hernia repair

SECONDARY OUTCOMES:
Effect of IPSS | 2 weeks
  the variance in the relationship between treatment arm and incidence of post-operative urinary retention in patients undergoing hernia repair that is attributable to International Prostate Symptom Score (IPSS)

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Health University Medical Center, Savannah, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.